CLINICAL TRIAL: NCT06089746
Title: Lumbosacral Spinal Stenosis - Non-Invasive Postural Therapy for Older Adult Veterans (LSS-NIPT)
Brief Title: Lumbosacral Spinal Stenosis - Non-Invasive Postural Therapy for Older Adult Veterans
Acronym: LSS-NIPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: E4412-P
Record Dates: First submitted 2023-08-21; First posted 2023-10-18 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — dichlorobis(azomycin)platinum II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Feasibility (Experimental): Patients with LSS will receive DME and training to support continuous maintenance of flexion posture during the 6 week trial. All participants will be asked to wear actigraphs and pedometers intermittently and to complete questionnaires and mobility assessments.
  Interventions: Other: NIPT

INTERVENTIONS:
Other: NIPT — Coordinated suite of DME and training to support continuous maintenance of flexion posture during the 6 week trial.

SUMMARY:
Lumbosacral spinal stenosis (LSS) is a leading cause of limited mobility, reduced independence, and poor health outcomes in older adults, and is very common in older adult Veterans. Several years ago, major research studies indicated that surgery for LSS was more effective than usual (medical) management. Nonetheless, there are many patients for whom surgery is not the ideal therapy. There have been reports that modifications in daily activities including temporary use of a modified rolling walker and changes in sleep positioning may help relieve LSS. The investigators have assembled a VA team to study this carefully. The investigators will recruit a small group of older adult Veterans with LSS to try out this program; the investigators will monitor them closely for relief of their symptoms and improvements in walking. The investigators will, as part of this small study, try to understand potential barriers to use of this therapy. The investigators will interview the Veterans and healthcare providers to identify problems that may arise in trying this therapy. If this small study works, the investigators plan to expand the effort.

ELIGIBILITY:
Inclusion Criteria:

* Veterans receiving care at participating VA
* Ability to read and write English and understand instructions
* Agrees to comply with instructions
* Symptoms for over 3 months
* Diagnosis of Lumbar Spinal Stenosis as the cause of symptoms
* Discomfort involving low back pain and / or neurogenic claudication of legs or thighs
* Back and/or leg symptoms greater than 3/10 provoked by walking and / or standing
* X ray, CT, or MRI performed within the last 12 months shows Lumbar Spinal Stenosis at 1 or 2 levels
* Prior treatment for Spinal Stenosis including therapy, medication, epidural injections, but not surgery
* Relief of pain (standardly within 5 minutes) by sitting down
* Ability to walk 50 feet without a cane or walker
* General health presents ability to increase activity level if Back and / or leg symptoms resolve
* If home has stairs and patient uses multiple levels, must have steady handrail
* Transportation routinely available by car or car service and not by bus
* Home location allows restriction of walking to flat surfaces (lack of hills), with availability to increase ambulation on flat surfaces

Exclusion Criteria:

* Previous Low Back Surgery for SS including decompression or fusion
* Successful Spinal Stenosis Treatment (such as injection) over the prior 3 months
* X ray, CT, or MRI shows Lumbar Spinal Stenosis in 3 or 4 levels
* Prior Lumbar Fracture
* Scoliosis with Cobb angle over 20 degrees on weight bearing AP Views
* Inflammatory arthropathy involving the Lumbar Spine, such as RA
* Radiculopathy attributed to herniated disc
* Suspected or confirmed moderate to severe large fiber neuropathy
* Failure of relief of back or leg pain brought on by standing or walking, within 5 minutes, by sitting down
* Rapid increase in symptoms with lumbar flexion such as sitting, Increase in symptoms brought on by leaning on grocery cart or walker
* Reduced symptoms by lumbo-sacral extension
* Vascular Claudication with ABI less than 60 or over 140
* Prior bypass or stent surgery for PAD
* Current foot, ankle, leg, or thigh infection or open ulcer
* Current use of a Brace for foot, ankle, or knee pathology,
* Moderate to severe arthritis of the Hip, knee, ankle or foot preventing pain free ambulation greater than 1 block
* Neurologic or neurodegenerative induced gait pathology such as CVA, Parkinson's, NPH, Cervical Myelopathy
* Current Medico Legal issues, active substance use, SI, HI, or other factors that may interfere with completion of six-week treatment trial
* Planned surgery or procedure in the 6-week study period

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in mobility by actigraph (positive, negative, or zero) as determined by the difference in mobility at Week 6 compared to baseline | Week 6
  Actigraph mobility

CONTACTS AND LOCATIONS:
Overall Officials: Beth B. Hogans, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset will be created and shared pursuant to a Data Use Agreement appropriately limiting the use of the dataset and prohibiting the recipient from identifying or re-identifying or taking steps to identify or re-identify any individual whose data are included in the dataset.